CLINICAL TRIAL: NCT02958761
Title: Treatment of Knee Arthrosis: Platelet-derived Growth Factors vs. Hyaluronic Acid. A Phase II-III Randomized Controlled Trial
Brief Title: Treatment of Knee Arthrosis With Platelet-derived Growth Factors vs. Hyaluronic Acid.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Claudio Lisi, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28914/2009
Record Dates: First submitted 2016-10-29; First posted 2016-11-08 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Knee Osteoarthrosis
Keywords: knee arthrosis; platelet-derived growth factors
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Platelet-rich plasma (Experimental): Patients in the intervention group will receive three autologous PRP plus calcium gluconate (as activator) intraarticular injections at 4-week intervals. Briefly, at the Immunohaematology and Transfusion Service, on each scheduled visit 20 ml of autologous whole blood will be sampled from each patient, 2 ml ACD-A will be added directly the syringe as anticoagulant; finally the vial will be gently centrifuged at 900rpm for 7 minutes. Platelet-rich plasma was collected. The PRP vials plus activator will be immediately shipped to the rehabilitation unit, where intraarticular injection will be performed by an experienced physiatrist.
  Interventions: Biological: intraarticular injections of platelet lysate
- hyaluronic acid (Active Comparator): Patients in the control group will receive three intraarticular hyaluronic acid (20 mg/2 mL; Hyalgan, Fidia, Abano Terme, Italy) injections at the same intervals, by the same study staff.
  Interventions: Drug: hyaluronic acid

INTERVENTIONS:
Biological: intraarticular injections of platelet lysate
  Arms: Platelet-rich plasma
Drug: hyaluronic acid — intraarticular hyaluronic acid (20 mg/2 mL; Hyalgan, Fidia, Abano Terme, Italy) injections at the same intervals
  Arms: hyaluronic acid

SUMMARY:
Primary aim of this trial was to assess efficacy three intraarticular injections of platelet lysate when compared to hyaluronic acid. Additional objectives were to compare the treatment groups in terms of a number of functional scales and of number of adverse events.

DETAILED DESCRIPTION:
Intra-articular injections of hyaluronic acid are effective in improving symptoms and slow disease progression, but are not able to revert the damage mechanism and trigger cartilage healing.

Growth factors included in PRP could stimulate cartilage repair, normalize synovial fluid viscoelasticity, induce a correction in tissue damage, improve articular function, control pain and ameliorate quality of life.

Primary aim of this trial was to assess, among patients with grade II/III osteoarthrosis of the knee, efficacy (as determined by improvement at MRI 6 months after the first injection) of three intraarticular injections of platelet lysate when compared to hyaluronic acid. Additional objectives were to compare the treatment groups in terms of a number of functional scales (WOMAC, Lysholm, Tegner Knee, Scale, AKS, Lequesne, VAS) and of number of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* grade II/III OA of the knee demonstrated at MRI17,18, according to Shahriaree Classification System - modified
* no previous OA treatment with local hyaluronic acid or steroid injections
* ife expectancy >1 year
* no ongoing pregnancy
* ability to understand and complete clinical and functional scales Lysholm, WOMAC, AKS, VAS
* written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-08; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Efficacy (as determined by improvement at MRI 6 months after the first injection) of intraarticular injections of platelet lysate | Six months after the last infiltration
  Each knee was improvement, from baseline, by at least one degree the maximum MRI score (Shahriaree Classification System - modified) at 6 month

SECONDARY OUTCOMES:
WOMAC functional scale | At baseline (prior to treatment), at 15 days form the last injection, 6 months from the last infiltration and at 1 year
  multilevel generalized linear models (for panel-data) with interaction between time and treatment group
Lysholm functional scale | At baseline (prior to treatment), at 15 days form the last injection, 6 months from the last infiltration and at 1 year
  multilevel generalized linear models (for panel-data) with interaction between time and treatment group
Tegner Knee functional scale | At baseline (prior to treatment), at 15 days form the last injection, 6 months from the last infiltration and at 1 year
  multilevel generalized linear models (for panel-data) with interaction between time and treatment group
AKS functional scale | At baseline (prior to treatment), at 15 days form the last injection, 6 months from the last infiltration and at 1 year
  multilevel generalized linear models (for panel-data) with interaction between time and treatment group
Lequesne functional scale | At baseline (prior to treatment), at 15 days form the last injection, 6 months from the last infiltration and at 1 year
  multilevel generalized linear models (for panel-data) with interaction between time and treatment group
VAS for pain | At baseline (prior to treatment), at 15 days form the last injection, 6 months from the last infiltration and at 1 year
  multilevel generalized linear models (for panel-data) with interaction between time and treatment group
Adverse event | 1 year
  number of patients and knees with adverse event (any); anticipated potential adverse events were infection, anaphylaxis, hematoma

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Lisi, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia

IPD SHARING:
Plan to Share IPD: No